CLINICAL TRIAL: NCT03591042
Title: Universal Transvaginal Cervical Length Screening Program for Prevention of Preterm Birth in Singletons Without Prior Preterm Birth: a Randomized Controlled Trial
Brief Title: Universal Transvaginal Cervical Length Screening Program for Prevention of Preterm Birth in Singletons Without Prior Preterm Birth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 31/18
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical length screening (Experimental): cervical length screening
  Interventions: Diagnostic Test: cervical length screening
- no screening (No Intervention): no screening

INTERVENTIONS:
Diagnostic Test: cervical length screening — transvaginal ultrasound cervical length
  Arms: cervical length screening

SUMMARY:
This is a non-blinded randomized screening trial of asymptomatic singleton pregnancies without prior spontaneous preterm birth who are randomized to either transvaginal ultrasound cervical length screening program (i.e. intervention group) or no screening (i.e. control group). Women are consented and randomized at the time of their routine anatomy scan between 18 0/7 and 23 6/7 weeks. Women randomized in the transvaginal ultrasound cervical length screening will receive a single transvaginal ultrasound cervical length measurement after the anatomy scan. The cervical length will be measured by operators with certification of competence in the technique.

ELIGIBILITY:
Inclusion criteria are:

* Singleton gestations
* No prior SPTB

Exclusion criteria are:

* Multiple gestations
* History of SPTB in a prior pregnancy
* Rupture of membranes at the time of randomization
* Known major fetal structural (i.e. defined as those that are lethal or require prenatal or postnatal surgery) or chromosomal abnormality
* Fetal death at the time of randomization
* Cerclage in situ at the time of randomization
* Pessary in situ at the time of randomization
* Vaginal bleeding at the time of randomization
* Women who are unconscious, severly ill, mentally handicapped, or under the age of 18 years.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 1334 (Estimated)
Dates: Start 2018-07-21 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
preterm birth rate | Less than 37 weeks
  either spontaneous or indicated preterm delivery

SECONDARY OUTCOMES:
preterm birth rate | ess than 24, 28, 32, 30, and 34 weeks gestation
  either spontaneous or indicated preterm delivery
admission to neonatal intensive care unit | time of delivery
neonatal death | Between birth and 28 days of age
birth weight | time of delivery
  weight of the baby at the time of delivery
Composite of adverse perinatal outcomes | Between birth and 28 days of age
  Number of neonates who will have at least one of the following: necrotizing enterocolitis (NEC), intraventricular hemorrhage (IVH) (grade 3 or higher), respiratory distress syndrome (RDS), bronchopulmonary dysplasia (BPD), retinopathy (ROP), blood-culture proven sepsis and neonatal death
perinatal death | Between birth and 28 days of age
  either fetal or neonatal mortality

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Gabriele Saccone, Naples
  - Seconda Università di Napoli Luigi Vanvitelli, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saccone G, Maruotti GM, Morlando M, Visentin S, De Angelis C, Sarno L, Cosmi E, Torcia F, Costanzi F, Gragnano E, Bartolini G, La Verde M, Borelli F, Savoia F, Schiattarella A, De Franciscis P, Locci M, Guida M; Italian Preterm Birth Prevention (IPP) Working Group. Randomized trial of screening for preterm birth in low-risk women - the preterm birth screening study. Am J Obstet Gynecol MFM. 2024 May;6(5S):101267. doi: 10.1016/j.ajogmf.2023.101267. Epub 2024 Feb 19. PMID 38642994